CLINICAL TRIAL: NCT01505725
Title: Nicotine Reinforcement and Smoking-Cue Reactivity: Association With Genetic Polymorphisms
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910456; 10-DA-N456
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-11-29

CONDITIONS: Nicotine Dependence
Keywords: Nicotine Reinforcement; Tobacco Craving; Behavior Genetics; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Researchers have been studying behavioral components of nicotine addiction by looking at how drugs have a reinforcing effect, connecting the stimulation provided by the drug (nicotine) to the behavior that produces it (smoking). Based on previous studies, researchers are interested in learning more about how nicotine affects current smokers' responses to psychological tests and smoking-related cues, and in studying whether certain kinds of genetic background may affect smokers' responses to these kinds of studies.

Objectives:

* To compare the effect of nicotine versus denicotinized cigarettes during specific psychological tests.
* To compare the effects of smoking cues versus neutral cues on craving, mood, and autonomic response.
* To study the effect of genes on nicotine reinforcement and smoking-cue reactivity.

Eligibility:

- Individuals between 18 and 64 years of age who are current smokers (at least 10 cigarettes per day for at least 1 year) and are not currently interested in reducing their smoking or seeking treatment for tobacco dependence.

Design:

* Pilot session:
* Participants will practice smoking using the measuring equipment that will be used in the study.
* After successful practice, participants will read or listen to music for 1 hour, during which they are not allowed to smoke.
* After the 1-hour period, participants will sample study cigarettes that have different levels of nicotine, and will be asked to guess whether the cigarettes are normal study cigarettes or denicotinized cigarettes.
* Baseline session:
* Blood, urine, and breath samples will be taken at the start of the session.
* Participants will smoke part of an initial cigarette, and then will read or listen to music for 1 hour, during which they are not allowed to smoke.
* After the 1-hour period, participants will give another breath sample and will complete questionnaires about mood and concentration levels.
* Trial sessions:
* Participants will smoke study cigarettes, and will be asked to either respond to questions about perceived nicotine levels in the cigarettes or press a lever for the chance to be rewarded with additional puffs of the cigarette. After the session, participants will give another breath sample and will complete questionnaires about mood and concentration levels.
* Participants will also participate in cue-reactivity sessions to test the body's physiological response to smoking cues (a pack of cigarettes) and neutral cues (a pack of unsharpened pencils). After the session, participants will complete questionnaires on mood and concentration 15, 30, 45, and 60 minutes after the session.
* At the conclusion of the last experimental session, participants will discuss the study with researchers, and may receive a referral list of smoking treatment programs.

DETAILED DESCRIPTION:
Objectives: 1) to compare the reinforcing efficacy of nicotine versus denicotinized cigarettes using a forced choice and an operant response procedure, 2) to compare the effects of smoking cues versus neutral cues on craving, mood, and autonomic responsivity, and 3) to explore potential associations between several genetic polymorphisms and the phenotypic measures of nicotine reinforcement and smoking-cue reactivity.

Study population: 175 adult smokers (35 for pilot study I, 60 for pilot stufy II and 80 for main study).

Design: Placebo-controlled, within-subjects design. Pilot studies will entail 1-2 sessions. Main study will entail one baseline/adaptation session and 5-10 experimental sessions.

Outcome Measures:

Behavioral Measures

During forced-choice sessions, primary measure is the percentage of nicotine cigarette puffs chosen and taken during choice trials. During operant response sessions, primary measures include breakpoint (final ratio completed), total number of responses, and number of cigarette puffs earned and taken. During cue-reactivity sessions, primary measures include craving, mood, and autonomic responsivity (heart rate, blood pressure, skin conductance, and skin temperature).

Genetic Measures

The following genetic polymorphisms will be assayed: 1) C/T rs2023239 variant of the CB1R gene, 2) the Ser/Gly rs6280 variant of DRD3 gene, and 3) variants of the CYP2A6 gene.

Secondary Measures

Secondary study measures include baseline smoking history, FTND, TCQ-SF, mood form, CO, and urinary cotinine and 3-hydroxycotinine. The ratio of 3-hydroxycotinine/cotinine is a phenotypic biomarker of the rate of nicotine metabolism, which has been shown to be associated with CYP2A6 genotype, level of nicotine dependence, various smoking behaviors, and treatment outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18-64 year old males and females
  2. smoking at least 10 cigarettes per day for at least 1 year
  3. urinary cotinine level greater than or equal to 100 ng/ml (NicAlert reading greater than or equal to 3)
  4. medically and psychologically healthy as determined by screening criteria

EXCLUSION CRITERIA:

1. definite plan to reduce or quit tobacco use in the next 30 days
2. treatment for tobacco dependence in the past 3 months
3. use of nicotine replacement products, bupropion, or varenicline in the past 3 months
4. consumption of more than 15 alcoholic drinks per week during the past month
5. use of any illicit drug more than twice per week during the past month
6. current use of any medication that would interfere with the protocol in the opinion of MAI
7. under the influence of a drug or alcohol at experimental sessions
8. pregnant, nursing, or become pregnant during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2010-03-16; Study Completion 2013-11-29

PRIMARY OUTCOMES:
Choice of nicotine cigarettes; cue-elicited craving

SECONDARY OUTCOMES:
smoking history measures; variants of several genes related to nicotine additions

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Bickel WK, Hughes JR, DeGrandpre RJ, Higgins ST, Rizzuto P. Behavioral economics of drug self-administration. IV. The effects of response requirement on the consumption of and interaction between concurrently available coffee and cigarettes. Psychopharmacology (Berl). 1992;107(2-3):211-6. doi: 10.1007/BF02245139. PMID 1615122
- [Background] Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory factor analyses and reliability of the modified cigarette evaluation questionnaire. Addict Behav. 2007 May;32(5):912-23. doi: 10.1016/j.addbeh.2006.06.028. Epub 2006 Jul 27. PMID 16875787
- [Background] Carter BL, Tiffany ST. Meta-analysis of cue-reactivity in addiction research. Addiction. 1999 Mar;94(3):327-40. PMID 10605857